CLINICAL TRIAL: NCT04846335
Title: Familiar Fatal Insomnia: Preventive Treatment With Doxycycline in Subject With Disease Risk
Acronym: FFI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Collaborators: Fondazione Telethon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FFI
Record Dates: First submitted 2021-04-12; First posted 2021-04-15 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2021-04

CONDITIONS: Familial Fatal Insomnia
MeSH Terms: conditions — Insomnia, Fatal Familial

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The protocol provided that in the trial were included carriers and non-carriers, members of the FFI family, who followed exactly the same procedures with the only difference that non-carriers received the placebo instead of the DOXY, since we could not exclude that a participant, by accidentally discovering that he/she received DOXY, automatically would realize to belong to the carrier group, we decided that also the non-carrier people will receive DOXY with a random schedule for a limited period of time so to eliminate any possible association. Only study coordinator will be informed about the presence of the mutation and will perform drug allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Bassado (Experimental): patients with D178N/M129 mutation on prion protein will be treated with Bassad
  Interventions: Drug: Doxycycline Hcl
- Placebo (Placebo Comparator): subject without the mutation will be treated with plac
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Doxycycline Hcl — tablets of DOXY hydrocloride (Bassado)
  Arms: Active Bassado
Drug: Placebo — tablets of placebo
  Arms: Placebo

SUMMARY:
The neurodegenerative disorders is a class o pathologies including very common diseases as Alzheimer or Parkinson or very rare as fatal familial insomnia (FFI), the progression of the disease with no therapeutic remedy is the common tract of these disorders. The aim of this project is to carry out a preventive treatment in subjects with genetic risk to develop FFI to avoid the establishment of the disease. FFI is a rare genetic neurodegenerative disease characterized by disrupted sleep, autonomic hyperactivation and motor abnormalities with fatal exitus. FFI is inherited in an autosomal dominant fashion and is linked to the D178N mutation in the prion protein gene (PRNP) in association with a methionine at the polymorphic codon 129 (D178N/M129). About thirty FFI pedigrees have been described worldwide, the mfirst case being reported in 1986 in northern Italy. This patient turned out to belong to large kindred, which spans 7 generations dating back to the eighteenth century. Many people belonging to this geneaology still live in the Veneto region of Italy, and they are part of an association. The genetic screening of 85 subjects belonging to this family permitted to identify the mutation carriers. Since the disease is aggressive and the affected people usually died within thirteen months from the onset, the possibility of an efficacious therapy when the disease become evident is unrealistic. This condition indicates in a preventive approach the better condition to affect the disease. Experimental studies and clinical observation indicated the antibiotic doxycycline (DOXY) as a potential candidate for a treatment in FFI subjects. The age with maximal risk to get the disease is between 50 and 55 years old. Thus the carriers that were born between 1958 and 1969 will be recruited for a preventive treatment with DOXY for ten years, at the end of this period or before we can establish if DOXY can be useful to avoid the development of FFI.

ELIGIBILITY:
Inclusion Criteria:

* subjects aged 44 to 53 years;
* no conditions known to be contraindications to the use of tetracyclines;
* written informed consent.

Exclusion Criteria:

* end stage liver,
* heart and renal disease,
* active malignancy,
* female subjects who are pregnant or lactating

Ages: 44 Years to 53 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2011-04-28 (Actual); Primary Completion 2021-04-12 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
survival | after 10 years of treatment
  The efficacy of the preventive treatment will be evaluated on the percentage of the survivals after ten years, according to the statistical analysis if no more than three individuals will die within the ten years, the treatment can be considered active to prevent FFI insurgence.

IPD SHARING:
Plan to Share IPD: No